CLINICAL TRIAL: NCT02659514
Title: A Phase 2 Study of Poziotinib in Patients With HER2-Positive Metastatic Breast Cancer (MBC) Who Have Received Prior HER2 Regimens for MBC
Brief Title: Study of Poziotinib in Participants With HER2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-201
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Poziotinib; Metastatic Breast Cancer; HER2-positive; Pan-HER inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Poziotinib 24 mg (Experimental): Participants received poziotinib 24 milligrams (mg), administered as three 8 mg tablets, orally, once daily (QD) on an intermittent dosing schedule of 14 days on treatment followed by 7 days off treatment, in a 21-day cycle until disease progression, death, intolerable adverse events (AEs) or for up to a maximum of 24 months, whichever occurs first.
  Interventions: Drug: Poziotinib
- Cohort 2: Poziotinib 16 mg (Experimental): Participants received poziotinib 16 mg, administered as two 8 mg tablets, orally, QD, on a continuous dosing schedule in a 21-day cycle until disease progression, death, intolerable AEs or for up to a maximum of 24 months, whichever occurs first.
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — 8 mg oral tablets, administered QD.
  Other Names: HM781-36B

SUMMARY:
The purpose of this study is to establish the dose regimen and evaluate the preliminary efficacy and the safety/tolerability of poziotinib in participants with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer who have received at least two prior HER2-directed treatment regimens.

DETAILED DESCRIPTION:
This is a phase 2, open-label, multicenter study to establish the dose regimen and evaluate the preliminary efficacy and the safety/tolerability of poziotinib in participants with HER2-positive metastatic breast cancer who have received at least two prior HER2-directed treatment regimens.

Each treatment cycle will be 21 days in duration. During each 21-day cycle, participants who are eligible for participation will receive poziotinib orally once daily.

All treated participants will be followed up until disease progression, death, intolerable adverse events or up to a maximum of 24 months whichever comes earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed primary breast cancer with metastatic lesions.
2. Confirmed HER2 overexpression or gene-amplified tumor
3. At least two prior HER2-directed therapy regimens for breast cancer, including trastuzumab and trastuzumab emtansine
4. Measurable disease per Response Evaluation Criteria for Solid Tumors version 1.1 (RECIST v1.1)
5. Participant is at least 18, and ≤90 years of age.
6. Adequate hematologic, hepatic, and renal function
7. Eastern Cooperative Oncology Group (ECOG) performance status <= 2

Exclusion Criteria:

1. Previous treatment with poziotinib prior to study participation
2. Brain metastases that are symptomatic or require therapy to control symptoms, as well as any history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 15 days of enrollment.
3. Anticancer chemotherapy, biologics, immunotherapy, cure-intent radiotherapy, or investigational treatment within 15 days, except for hormone therapy, palliative therapy, or supportive therapy.
4. History of congestive heart failure Class III/IV according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment.
5. Cardiac ejection fraction <50%
6. History of other malignancies within the last 5 years
7. Participant is pregnant or breast-feeding.
8. Unable to take drugs orally

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (35):
- United States (35):
  - Clearview Cancer Center, Huntsville, Alabama
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Marin Cancer Care, Inc, Greenbrae, California
  - Alliance Research Centers, Laguna Hills, California
  - PacificShores Medical Group, Long Beach, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Innovative Clinical Research Institute, Whittier, California
  - AMPM Research Clinic, Miami Gardens, Florida
  - FL Cancer Research Institute, Plantation, Florida
  - Bond Clinic, P.A., Winter Haven, Florida
  - Triple Army Medical Cente, Honolulu, Hawaii
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Hattiesburg Clinic Hematology Oncology, Hattiesburg, Mississippi
  - Washington University, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - White Plain Hospital, White Plains, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma Cancer Specialists & Research Institute, LLC, Tulsa, Oklahoma
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Oncology Consultants, P.A., Houston, Texas
  - SAMMC - Hem/Onc Clinic, Houston, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Providence Regional Cancer System, Lacey, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 participants were enrolled at 19 sites in the United States in the study which was conducted from 22 February 2016 to 11 March 2020.
Period: Overall Study
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Started | 33 | 34
Safety Population (Safety Population included all participants who received at least one dose of poziotinib.) | 33 | 34
Evaluable Population (Evaluable Population included all participants who had received at least one cycle of poziotinib and had at least one evaluable post-baseline tumor response evaluation using response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST, v1.1).) | 30 | 27
Completed | 1 | 0
Not Completed | 32 | 34
Not completed — Adverse Event | 3 | 12
Not completed — Disease Progression | 23 | 13
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 6 | 1
Not completed — Reason Unspecified | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of poziotinib.
Groups:
- Cohort 1: Poziotinib 24 mg: Participants received poziotinib 24 mg, administered as three 8 mg tablets, orally, QD on an intermittent dosing schedule of 14 days on treatment followed by 7 days off treatment, in a 21-day cycle until disease progression, death, intolerable AEs or for up to a maximum of 24 months, whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (13.82) | 58.1 (11.10) | 57.3 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response (BOR) was complete response (CR) or partial response (PR) among participants in the Evaluable Population assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). ORR was based on investigator assessed BOR. Per RECIST v1.1 for target lesions, CR was disappearance of all target tumor lesions (TLs) and all target lymph nodes (LNs) with short axis <10mm. PR was ≥30% decrease in sum of diameters (SOD) from Baseline, and not progressive disease (PD) (≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm).
Time Frame: Up to 24 months
Population: Evaluable Population included all enrolled participants who completed at least 1 cycle of poziotinib treatment and had at least 1 post-baseline tumor response evaluation using RECIST, v 1.1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 30 | 27
percentage of participants | 30 [14.7 to 49.4] | 30 [13.8 to 50.2]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was the duration of time (in months) from first administration of study treatment to date of first documented disease progression or death from any cause. PFS of living participants without documented PD was censored at the time of last tumor assessment or the date of first treatment if there was no post-baseline tumor assessment. Per RECIST v1.1 for target lesions, PD was defined as ≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm.
Time Frame: Up to 24 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 30 | 27
months | 4.1 [1.5 to 5.6] | 4.9 [1.8 to 7.4]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was the percentage of participants whose best response was CR, PR or stable disease (SD) among participants in the Evaluable Population assessed per RECIST v1.1. DCR was based on investigator-assessed BOR. Per RECIST v1.1 for target lesions, CR was defined as disappearance of all target TLs and all target LNs with short axis <10mm. PR was ≥30% decrease in sum of diameters (SOD) from Baseline, and not progressive disease (≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm). SD was SOD change neither sufficient for PR nor sufficient for PD.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 30 | 27
percentage of participants | 60 [40.6 to 77.3] | 78 [57.7 to 91.4]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time (in months) from first administration of study drug to tumor progression, which excluded death without tumor progression, by the end of study. TTP of participants who died without documented PD was censored at date of death. TTP of living participants without documented PD was censored at the same time as PFS, which was the last tumor assessment or the date of first treatment if there was no post-baseline tumor assessment. Per RECIST v1.1 for target lesions, PD was defined as ≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 30 | 27
months | 4.1 [1.5 to 5.6] | 4.9 [1.8 to 7.4]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR was evaluated only for participants whose BOR was CR or PR and was defined as the time (in months) from the date that response evaluation criteria were first met for CR or PR (whichever status was recorded first) until the first subsequent date that PD or death was documented. DoR of participants without documented PD or death was censored at the time of last tumor assessment. Per RECIST v1.1 for target lesions, CR was defined as disappearance of all target tumor lesions (TLs) and all target lymph nodes (LNs) with short axis <10mm. PR was defined as ≥30% decrease in sum of diameters (SOD) from Baseline, and not PD. PD was defined as ≥20% increase in SOD from previous smallest SOD on study, and an absolute increase of ≥5mm).
Time Frame: Up to 24 months
Population: Evaluable Population included all participants who had received at least one cycle of poziotinib and had at least one evaluable post-baseline tumor response evaluation using response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST, v1.1). Overall number of participants analyzed is the number of participants with best overall response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 9 | 8
months | 5.7 [1.8 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with event. | 13.0 [2.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event.

6. Secondary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were AEs that occurred or worsened from the first dose of study treatment until 35 (± 5) days after the last dose of study treatment.
Time Frame: From the first dose of study drug administration until 35 (± 5) days after the last dose of study drug administration (Up to approximately 25 months)
Population: Safety Population included all participants who received at least 1 dose of poziotinib.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 33 | 34
participants | 33 | 33

7. Secondary Outcome: Pharmacokinetic Analysis (Drug Concentration Measurements)
Time Frame: For Cohort 1: Pre-dose and 1 and 2 hours post-dose on Day 1 of Cycles 1, 2, and 3, and pre-dose on Day 14 of Cycle 1 For Cohort 2: Day 1 of Cycle 1 pre-dose and 30 minutes, 1,1.5,2,3, 4, 6, and 24 hours post-dose of Day 1 of Cycle 1
Population: Pharmacokinetic analyses specified in the protocol were not performed as the samples were no longer stable at the time of the analysis.
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From the first dose of study drug administration up to approximately 48.5 months; Serious and Other Adverse Events: From the first dose of study drug administration until 35 (± 5) days after the last dose of study drug administration (up to approximately 25 months)
Description: Safety population included all participants who received at least 1 dose of poziotinib.
Arm/Group | Cohort 1: Poziotinib 24 mg | Cohort 2: Poziotinib 16 mg
All-Cause Mortality (participants affected / at risk) | 6/33 | 1/34
Serious Adverse Events (participants affected / at risk) | 14/33 | 16/34
Other Adverse Events (participants affected / at risk) | 33/33 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Poziotinib 24 mg (N=33) | Cohort 2: Poziotinib 16 mg (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Poziotinib 24 mg (N=33) | Cohort 2: Poziotinib 16 mg (N=34)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 1
Eye discharge (Eye disorders) | 2 | 1
Cataract (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 30 | 29
Stomatitis (Gastrointestinal disorders) | 16 | 17
Vomiting (Gastrointestinal disorders) | 16 | 11
Nausea (Gastrointestinal disorders) | 12 | 17
Constipation (Gastrointestinal disorders) | 5 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 18 | 17
Mucosal inflammation (General disorders) | 8 | 5
Pyrexia (General disorders) | 4 | 5
Oedema peripheral (General disorders) | 4 | 3
Pain (General disorders) | 4 | 1
Asthenia (General disorders) | 2 | 2
Chills (General disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 3
Oedema (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Infusion site rash (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Tenderness (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 1
Paronychia (Infections and infestations) | 4 | 3
Conjunctivitis (Infections and infestations) | 3 | 0
Fungal infection (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Rash pustular (Infections and infestations) | 1 | 2
Candida infection (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Angular cheilitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1
Enterocolitis infection (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tongue fungal infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Nail injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 6 | 5
Blood creatinine increased (Investigations) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood potassium decreased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Blood uric acid increased (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 2
Lymphocyte count decreased (Investigations) | 1 | 2
White blood cell count increased (Investigations) | 1 | 2
Neutrophil count increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Glomerular filtration rate increased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Blood chloride decreased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 13 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 12
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 5 | 4
Dysgeusia (Nervous system disorders) | 3 | 4
Burning sensation (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 0
Agitation (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 20 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1
Koilonychia (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 3
Lymphoedema (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02659514/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02659514/SAP_001.pdf